CLINICAL TRIAL: NCT01868646
Title: Multicentre Double-blind Placebo-controlled Parallel-group Randomized Clinical Trial of Efficacy and Safety of Subetta in the Combined Treatment of Patients With Type II Diabetes Mellitus
Brief Title: Clinical Trial of Efficacy and Safety of Subetta in the Combined Treatment of Patients With Type II Diabetes Mellitus
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Materia Medica Holding (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: MMH-SU-004
Record Dates: First submitted 2013-05-27; First posted 2013-06-04 (Estimated); Results first posted 2019-03-04 (Actual); Last update posted 2019-05-31 (Actual); Status verified 2019-05

CONDITIONS: Type II Diabetes Mellitus
Keywords: Combined Treatment of Patients With Type II Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — subetta

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Subetta (Experimental)
  Interventions: Drug: Subetta
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Subetta — Each Subetta tablet contains a mixture of affinity purified polyclonal antibodies to β-subunit of the rINS (6 mg) and antibodies to eNOS (6 mg) in released-active form produced by the patented technology in accordance with the applicable European Pharmacopeia requirements.
  Standard therapy of type II diabetes mellitus + Subetta (1 tablet 4 times a day) for 36 weeks.
  Subetta: oral administration, per 1 intake - 1 tablet (keep in the mouth until complete dissolution, not at mealtime).
  Arms: Subetta
Drug: Placebo — Placebo (identical to Subetta in shape and taste tablet containing exсipients). Standard therapy of type II diabetes mellitus + Placebo (1 tablet 4 times a day) for 36 weeks.
  Placebo: oral administration, per 1 intake - 1 tablet (keep in the mouth until complete dissolution, not at mealtime).
  Arms: Placebo

SUMMARY:
The purpose of this study is:

* to assess clinical efficacy of Subetta in the combined treatment of type II diabetes mellitus;
* to assess safety of Subetta in the combined treatment of type II diabetes mellitus.

DETAILED DESCRIPTION:
Patients with type II diabetes mellitus are included in the trial. It is concerned those patients, who by the time of the trial receive basal insulin with metformin or metformin and sulfonylurea derivatives and with lack of optimal glycemic control (HbA1c>7.0%). For patients, which will be included in the trial (mainly middle aged patients without severe complications of diabetes), HbA1c>7.0% is the marker showing that optimal individual goal of glycemic control is not achieved.

If a patient meets inclusion criteria and does not show exclusion criteria he/she is randomized in one of 2 groups: Group 1 - the group receiving standard type II diabetes mellitus therapy + Subetta at a dose of 1 tablet 4 times a day; Group 2 - the group receiving standard type II diabetes mellitus therapy + Placebo under the regimen used for Subetta. The invented names of the drugs containing basal insulin, metformin and sulfonylurea derivatives used as standard type II diabetes mellitus therapy, should be unchanged for each patient during the whole trial.

All patients will receive glucometers and the appropriate glucose test strips, so they could self monitor blood glucose and register this data in their diaries.

The trial duration is 38 weeks; the main stages of the trial are conducted during screening, then in 4 weeks (Visit 2), in 12 weeks (Visit 3), in 24 weeks (Visit 4) and in 36 weeks (Visit 5). In 1 week after randomization and the onset of the trial therapy and between the visits to the study site (on weeks 8±1, 18±1and 30±1) an investigator collects data on patient's health and complaints (phone visits) to decide whether it is necessary to arrange unplanned visit to the site.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosed type II diabetes mellitus (according to WHO criteria, 1999 - 2006).
2. Patient's age from 18 to 65 years inclusive.
3. Level of glycosylated hemoglobin 7.0- 10.0 %.
4. Dose of basal insulin ≥10 units/day combined with metformin or with metformin and sulfonylurea derivatives during not less than 3 months prior to inclusion in the trial.
5. Body mass index ≥25.0 and ≤40.0kg/m^2.
6. Constant body weight (without fluctuations > 10% during not less than 3 months prior to inclusion in the trial).
7. Glomerular filtration rate ≥ 60 ml/ min/1.73m^2.
8. Stable dose of basal insulin for the last 3 months.(Permissible fluctuations are ±10%.)
9. Usage of contraceptive methods by both gender patients of reproductive age during the trial and within 30 days after ending the participation in the trial.
10. Availability of signed patient information sheet (Informed Consent form) for participation in the clinical trial.

Exclusion Criteria:

1. Acute diabetes mellitus complications for 3 months prior to inclusion in the trial (diabetic ketoacidosis, hyperosmolar hyperglycemic state, lacticemia, severe hypoglycemia and hypoglycemic coma).
2. Diabetic retinopathy, preproliferative, proliferative or terminal stages (based on the results of oculist examination during screening period or 6 months prior to the trial).
3. Diabetic nephropathy, proteinuria stage, chronic kidney disease on 3, 4 or 5 stage.
4. Diabetic microangiopathy:

   * ishemic heart disease (medical history of a sudden coronary death with successful reanimation, medical history of myocardial infarction, stable exertional angina III or IV FC; unstable angina; postinfarction cardiosclerosis; chronic heart failure III or IV FC);
   * cerebrovascular diseases (medical history of acute cerebrovascular accident; progressive vascular leukoencephalopathy; vascular dementia);
   * chronic obliterative peripheral vascular diseases (clinically significant);
   * diabetic neuroosteoarthropathy;
   * diabetic foot (clinically significant).
5. Heart rhythm disorder:

   * II-III atrioventricular block;
   * sick sinus syndrome;
   * long QT interval syndrome;
   * complete left bundle branch block;
   * block of 2/3 bundle branches;
   * WPW syndrome;
   * ventricular arrhythmia of III grade according Laun-Wolf;
   * paroxysmal supraventricular tachycardia;
   * paroxysmal/recurrent ventricular tachycardia;
   * atrial flutter and fibrillation;
   * ventricular flutter and fibrillation;
   * heart pacemaker implant.
6. Uncontrolled arterial hypertension characterized by the following blood tension values: systolic blood pressure over 160 mm Hg and/or diastolic blood pressure over 100 mm Hg.
7. Severe concomitant pathology including clinically significant cardio- vascular diseases of III - IV functional class (according to New York Heart Association classification, 1964), nervous and endocrine system diseases, including morbid obesity (body mass index≥40.0 kg/m^2), renal insufficiency, liver failure.
8. Medical history of pancreatectomy or transplantation of pancreatic/islet cells.
9. Medical history of renal transplantation.
10. Malignant neoplasms/suspected malignant neoplasms.
11. Exacerbations or decompensation of chronic diseases affecting a patient's ability to participate in the clinical trial.
12. The results of analysis of liver enzymes (alanine aminotransferase, aspartate aminotransferase) more than threefold exceeding of upper limit of normal values.
13. Level of fasting triglycerides >5.64 mmol/L.
14. Medical history of bariatric surgical operations.
15. Medical history of polyvalent allergy
16. Allergy/ intolerance to any of the components of medications used in the treatment.
17. Intake of medicines listed in the section "Prohibited concomitant treatment" for 3 months prior to the inclusion in the trial.
18. Pregnancy, breast-feeding.
19. Drug addiction, alcohol usage in the amount exceeding 2 units of alcohol per day.
20. Mental disorders of a patient.
21. Night work.
22. Participation in other clinical trials in the course of 3 months prior to the inclusion in the trial.
23. Patients, who from the investigator's point of view, will fail to comply with the observation requirements of the trial or with the intake regimen of the investigated medicines.
24. Other factors impeding patient's participation in the trial (for example, planned business trips or journeys).
25. Patient is related to the research personnel of the investigative site, who are directly involved in the trial or are the immediate relative of the researcher. The immediate relative includes husband/wife, parents, children or brothers (or sisters), regardless of whether they are natural or adopted.
26. Patient works for OOO "NPF "Materia Medica Holding" (i.e. is the company's employee, temporary contract worker or appointed official responsible for the carrying out the research) or the immediate relative.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 190 (Actual)
Dates: Start 2013-05-07 (Actual); Primary Completion 2016-06-15 (Actual); Study Completion 2016-06-15 (Actual)

CONTACTS AND LOCATIONS:
Locations (17):
- Russia (17):
  - State Healthcare Institution of Moscow "Central research institute of gastroenterology" of Department of health care of Moscow, Moscow
  - State Educational Institution of Higher Professional Education "Moscow State Medical Academy named after I.M. Sechenov", Moscow
  - Nonstate Health Care Institution "Central Clinical Hospital №2 named after N.A. Semashko of Public Limited Company "Russian Railways", Moscow
  - Municipal budgetary authority "Khimki Central Clinical Hospital", Moscow Region
  - Nizhny Novgorod regional State Budgetary Health Institution " Nizhny Novgorod regional Clinical Hospital named after N.A. Semashko ", Nizhny Novgorod Region
  - State Budgetary Educational Institution of High Professional Training "Rostov State Medical University" of Ministry of Health of Russian Federation, Department of Endocrinology, Rostov-on-Don
  - St. Petersburg State Budgetary Health Care Institution "City Polyclinic №6", Saint Petersburg
  - St. Petersburg State Budgetary Health Care Institution "City Polyclinic №77 of Nevsky District", The City Diabetes Center №4, Saint Petersburg
  - St. Petersburg State Budgetary Health Care Institution "Saint Venerable Martyr Elizaveta Municipal Hospital", Saint Petersburg
  - State Budgetary Educational Institution of High Professional Training "St. Petersburg State Medical University named after academician I.P. Pavlov" of Ministry of Health of Russian Federation, Therapy Faculty Board, Saint Petersburg
  - St. Petersburg Sate Budgetary Institution "Consultative-Diagnostic Polyclinic №1 of Coastal Area", Saint Petersburg
  - St. Petersburg State Budgetary Health Care Institution "Consultative-Diagnostic Center № 85", Diabetes Center №2, Saint Petersburg
  - Co.Ltd " Diabet Center", Samara
  - The State Budgetary Educational Institution of Higher Professional Education "Smolensk National Research Medical University" Ministry of Health of the Russian Federation, Smolensk
  - Vladimir region State budgetary institution of health care "Regional clinical hospital", Vladimir
  - Independent Health Care Institution of Voronezh Region "Voronezh Regional Clinical Consultative-Diagnostic Center", Voronezh
  - State Budgetary Health Care Institution of Yaroslavl Region "Regional Сlinical Hospital", Yaroslavl

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Selection procedures were carried out after participant enrollment to determine whether the patient could participate in the study in accordance with the inclusion/exclusion criteria.
  Of the 190 patients enrolled, 42 did not meet inclusion criteria after screening procedures, they were not randomized
Groups:
- Subetta: Standard therapy of type II diabetes mellitus + Subetta (1 tablet 4 times a day).
  Subetta: oral administration, per 1 intake - 1 tablet (keep in the mouth until complete dissolution, not at mealtime).
  One tablet contains: affinity purified antibodies to the C-terminal fragment of the beta subunit receptor insulin - 0.006g*, affinity purified antibodies to endothelial NO synthase - 0.006g*.
  *applied onto isomalt crystals as a mixture of three active aqueous-alcoholic dilutions of the drug substance - diluted 100^12, 100^30, 100^200 times, respectively.
  Excipients: isomalt, crospovidone, magnesium stearate.
- Placebo: Standard therapy of type II diabetes mellitus + Placebo (1 tablet 4 times a day).
  Placebo: oral administration, per 1 intake - 1 tablet (keep in the mouth until complete dissolution, not at mealtime).
  Placebo
Period: Overall Study
Arm/Group | Subetta | Placebo
Started | 76 | 72
Completed | 73 | 67
Not Completed | 3 | 5
Not completed — Do not meet inclusion criteria | 3 | 5

BASELINE CHARACTERISTICS:
Population: Intention-to-Treat set
Groups:
- Subetta: Standard therapy of type II diabetes mellitus + Subetta (1 tablet 4 times a day).
  Subetta: oral administration, per 1 intake - 1 tablet (keep in the mouth until complete dissolution, not at mealtime).
  Subetta: Efficacy and Safety of Subetta in the combined treatment of patients with type II diabetes mellitus
- Total: Total of all reporting groups
Arm/Group | Subetta | Placebo | Total
Number analyzed (Participants) | 73 | 67 | 140
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.9 (7.1) | 57.3 (6.2) | 57.6 (6.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 59 | 54 | 113
  Male | 14 | 13 | 27
Weight [Mean (Standard Deviation); unit: kilogram] | 85.7 (13.0) | 89.0 (11.7) | 87.1 (12.5)
Height [Mean (Standard Deviation); unit: centimeter] | 164.1 (7.7) | 165.3 (7.3) | 164.7 (7.5)
BMI [Mean (Standard Deviation); unit: kilogram/m^2] | 31.7 (4.0) | 32.5 (3.6) | 32.1 (3.8)

OUTCOME MEASURES:

1. Primary Outcome: Changes in the Mean Value of HbA1c
Description: The HbA1C test was performed using a method that is certified by the National Glycohemoglobin Standardization Program (NGSP) (www.ngsp.org) and standardized or traceable to the Diabetes Control and Complications Trial (DCCT) reference assay.
Time Frame: In 12, 24 and 36 weeks of the treatment as compared to the baseline
Population: Intention-to-Treat set
Measure: Mean (Standard Deviation); unit: percentage of HbA1c
Arm/Group | Subetta | Placebo
Number analyzed (Participants) | 73 | 67
percentage of HbA1c
  12 weeks | -0.53 (1.06) | -0.01 (1.06)
  24 weeks | -0.54 (1.00) | -0.07 (1.19)
  36 weeks | -0.54 (1.11) | 0.15 (1.07)
Statistical Analysis 1: Comparison: Subetta vs Placebo; Test type: Superiority; p = 0.0002, Mixed Models Analysis — The p-value associated with "treatment" factor of changes from baseline to Week 12, 24 and 36 endpoint between Subetta and Placebo treatment groups. Model includes treatment, visit and treatment*visit interaction

2. Secondary Outcome: Change in Fasting Plasma Glucose
Description: Based on the data of biochemical analysis
Time Frame: In 4, 12, 24 and 36 weeks of the treatment as compared to the baseline
Population: Intention-to-Threat set
Measure: Mean (Standard Deviation); unit: mmol / l
Arm/Group | Subetta | Placebo
Number analyzed (Participants) | 73 | 67
mmol / l
  4 weeks | -0.5 (2.6) | -0.1 (3.2)
  12 weeks | 0.0 (2.5) | 0.9 (3.3)
  24 weeks | 0.0 (2.9) | 0.9 (4.1)
  36 weeks | 0.0 (3.1) | 1.0 (3.7)
Statistical Analysis 1: Comparison: Subetta vs Placebo; Test type: Superiority; p = 0.0426, Mixed Models Analysis — The p-value associated with "treatment" factor of changes from baseline to Week 4, 12, 24 and 36 endpoint between Subetta and Placebo treatment groups. Model includes treatment, visit and treatment*visit interaction

3. Secondary Outcome: Change in Average Daily Blood Glucose From a 7-point Patient Self-monitoring of Blood Glucose (SMBG)
Description: A 7-point patient self-monitoring of blood glucose (SMBG): three measurements of blood glucose before the meal; three measurements of postprandial blood glucose (1-2 h after the start of the meal) and one measurement at 3:00 a.m.
Time Frame: During the whole study period (on weeks 4, 8, 12, 18, 24, 30 and 36 of the treatment) as compared to the baseline
Population: Intention-to-Treat set. The SMBG in 3 patients (2 in the Subetta and 1 in the Placebo) was excluded from the analysis due to mistakes in diaries.
Measure: Mean (Standard Deviation); unit: mmol / l
Arm/Group | Subetta | Placebo
Number analyzed (Participants) | 71 | 66
mmol / l
  4 weeks | -0.3 (1.5) | -0.5 (1.8)
  8 weeks | -0.3 (1.6) | -0.5 (1.7)
  12 weeks | -0.4 (1.7) | -0.4 (2.1)
  18 weeks | -0.2 (1.6) | -0.4 (1.6)
  24 weeks | -0.5 (1.6) | -0.5 (1.7)
  30 weeks | -0.3 (1.7) | -0.5 (1.5)
  36 weeks | -0.5 (1.9) | -0.6 (1.7)
Statistical Analysis 1: Comparison: Subetta vs Placebo; Test type: Superiority; p = 0.5990, Mixed Models Analysis — The p-value associated with "treatment" factor of changes from baseline to Week 4, 8, 12, 18, 24, 30 and 36 endpoint between Subetta and Placebo treatment groups. Model includes treatment, visit and treatment*visit interaction

4. Secondary Outcome: Mean Value of C-peptide
Description: Blood samples (for measurement of fasting plasma glucose, concentrations of plasma C-peptide, total cholesterol, HDL cholesterol, LDL cholesterol and triglycerides) are taken under standard conditions: after night break in food taking (at least 8 hours) and prior to administering of insulin morning dose (if patient receives intermediate insulin twice-daily), prior to any morning medicines intake (including the study drug, metformin, sulfonylurea derivatives, permitted concomitant therapy).
Time Frame: In 12, 24 and 36 weeks of the treatment as compared to the baseline
Population: Intention-to-Treat set.
Measure: Mean (Standard Deviation); unit: pmol / l
Arm/Group | Subetta | Placebo
Number analyzed (Participants) | 73 | 67
pmol / l
  0 week | 615.3 (418.9) | 607.6 (425.4)
  12 weeks | 628.3 (400.8) | 607.7 (405.6)
  24 weeks | 643.3 (419.2) | 641.6 (426.3)
  36 weeks | 589.6 (343.5) | 540.0 (328.3)
Statistical Analysis 1: Comparison: Subetta vs Placebo; Test type: Superiority; p = 0.6215, Mixed Models Analysis — The p-value associated with "treatment" factor of mean value at baseline to Week 12, 24 and 36 endpoint between Subetta and Placebo treatment groups. Model includes treatment, visit and treatment*visit interaction

5. Secondary Outcome: Changes in Lipids (Concentrations of Plasma Total Cholesterol, HDL Cholesterol, LDL Cholesterol and Triglycerides)
Description: Blood samples (for measurement of fasting plasma glucose, concentrations of plasma total cholesterol, HDL cholesterol, LDL cholesterol and triglycerides) are taken under standard conditions: after night break in food taking (at least 12 hours) and prior to administering of insulin morning dose (prandial), prior to any morning medicines intake (including the study drug and permitted concomitant therapy).
Time Frame: In 12, 24 and 36 weeks of the treatment as compared to the baseline
Population: Intention-to-Treat set.
Measure: Mean (Standard Deviation); unit: mmol / l
Arm/Group | Subetta | Placebo
Number analyzed (Participants) | 73 | 67
mmol / l
  Total cholesterol (12 weeks) | 0.1 (1.1) | 0.1 (1.2)
  Total cholesterol (24 weeks) | 0.1 (1.2) | 0.1 (0.9)
  Total cholesterol (36 weeks) | 0.3 (1.1) | 0.0 (1.1)
  HDL cholesterol (12 weeks) | 0.0 (0.2) | 0.0 (0.2)
  HDL cholesterol (24 weeks) | 0.0 (0.2) | 0.0 (0.2)
  HDL cholesterol (36 weeks) | 0.0 (0.3) | 0.0 (0.2)
  LDL cholesterol (12 weeks) | 0.1 (0.8) | 0.0 (0.9)
  LDL cholesterol (24 weeks) | 0.1 (0.9) | 0.1 (0.8)
  LDL cholesterol (36 weeks) | 0.2 (0.8) | 0.1 (0.9)
  Triglycerides (12 weeks) | 0.2 (0.8) | 0.2 (0.9)
  Triglycerides (24 weeks) | 0.1 (0.9) | 0.0 (0.8)
  Triglycerides (36 weeks) | 0.1 (0.9) | -0.1 (0.9)
Statistical Analysis 1: Comparison: Subetta vs Placebo; Analysis of Total cholesterol changes from baseline to Week 12, 24 and 36 endpoint between Subetta and Placebo treatment groups; Test type: Superiority; p = 0.6155, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Subetta vs Placebo; Analysis of HDL cholesterol changes from baseline to Week 12, 24 and 36 endpoint between Subetta and Placebo treatment groups; Test type: Superiority; p = 0.7507, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Subetta vs Placebo; Analysis of LDL cholesterol changes from baseline to Week 12, 24 and 36 endpoint between Subetta and Placebo treatment groups; Test type: Superiority; p = 0.4195, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 4: Comparison: Subetta vs Placebo; Analysis of Triglycerides changes from baseline to Week 12, 24 and 36 endpoint between Subetta and Placebo treatment groups; Test type: Superiority; p = 0.3609, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]

6. Secondary Outcome: Changes in Dosage of Insulin (Basal Dose Insulin Measured in IU/Day)
Description: Changes in basal insulin dose is based on the mean value of 3 consecutive measuring of level of fasting blood glucose.
  1. If value of fasting blood glucose at 7:00 AM on January 21, 2012 - 4.2 mmol/L, at 7:30 AM on January 22, 2012- 5.0 mmol/L, at 7:00 AM on January 23, 2012 4.8 mmol/L, then the mean level of blood glucose =4.7 mmol/L (4.2 +5.0 +4.8 divided by 3). It is not recommended to change the dose.
  2. If the mean value of fasting blood glucose is lower than 4.0 mmol/L and a patient shows unreasonable signs or symptoms of hypoglycemia, then dose of basal insulin should be reduced by 2 units.
  3. If value of fasting blood glucose for 3 consecutive days was ≥7 mmol/L, then dose of basal insulin should be increased by 2 units and more (depending on individual values).
  Based on the same values investigator can change dose of per oral blood sugar-lowering drugs.
Time Frame: In 36 weeks of the treatment as compared to the baseline
Population: Intention-to-Treat
Measure: Mean (Standard Deviation); unit: IU/day
Arm/Group | Subetta | Placebo
Number analyzed (Participants) | 73 | 67
IU/day | -0.9 (2.4) | 3.5 (9.5)
Statistical Analysis 1: Comparison: Subetta vs Placebo; Test type: Superiority; p = 0.0605, t-test, 2 sided

7. Secondary Outcome: Changes in Dosage of Insulin (Basal Dose Insulin Measured in IU/ kg of Body Weight)
Description: Changes in basal insulin dose is based on the mean value of 3 consecutive measuring of level of fasting blood glucose.
  If value of fasting blood glucose at 7:00 AM on January 21, 2012 - 4.2 mmol/L, at 7:30 AM on January 22, 2012- 5.0 mmol/L, at 7:00 AM on January 23, 2012 4.8 mmol/L, then the mean level of blood glucose =4.7 mmol/L (4.2 +5.0 +4.8 divided by 3). It is not recommended to change the dose.
  If the mean value of fasting blood glucose is lower than 4.0 mmol/L and a patient shows unreasonable signs or symptoms of hypoglycemia, then dose of basal insulin should be reduced by 2 units.
  If value of fasting blood glucose for 3 consecutive days was ≥7 mmol/L, then dose of basal insulin should be increased by 2 units and more (depending on individual values).
  Based on the same values investigator can change dose of per oral blood sugar-lowering drugs.
Time Frame: In 36 weeks of the treatment as compared to the baseline
Population: Intention-to-Treat set
Measure: Mean (Standard Deviation); unit: IU/kg
Arm/Group | Subetta | Placebo
Number analyzed (Participants) | 73 | 67
IU/kg | -0.01 (0.03) | 0.04 (0.1)
Statistical Analysis 1: Comparison: Subetta vs Placebo; Test type: Superiority; p = 0.0726, t-test, 2 sided

8. Secondary Outcome: Percentage of Patients With Changed Daily Dose of Per Oral Blood Sugar- Lowering Drugs
Time Frame: In 36 weeks of the treatment
Population: Intention-to-Treat set
Measure: Number; unit: percentage of patients
Arm/Group | Subetta | Placebo
Number analyzed (Participants) | 73 | 67
percentage of patients | 4.1 | 9.0
Statistical Analysis 1: Comparison: Subetta vs Placebo; Test type: Superiority; p = 0.3108, Fisher Exact

9. Secondary Outcome: Changes in the Mean Absolute Value of Body Weight (kg)
Time Frame: In 36 weeks of the treatment as compared to the baseline
Population: Intention-to-Treat set. Data on body weight in one patient from the placebo group were absent
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Subetta | Placebo
Number analyzed (Participants) | 73 | 66
kg | -0.1 (2.2) | 0.4 (3.4)
Statistical Analysis 1: Comparison: Subetta vs Placebo; Test type: Superiority; p = 0.2934, t-test, 2 sided

10. Secondary Outcome: Changes in the Mean Absolute Value of Body Mass Index (BMI) (kg/m^2)
Time Frame: baseline and 36 weeks of the treatment
Population: Intention-to-Treat set. Data on body weight in one patient from the placebo group were absent
Measure: Mean (Standard Deviation); unit: kg/m^2
Arm/Group | Subetta | Placebo
Number analyzed (Participants) | 73 | 66
kg/m^2 | -0.04 (0.78) | 0.14 (1.33)
Statistical Analysis 1: Comparison: Subetta vs Placebo; Test type: Superiority; p = 0.3410, t-test, 2 sided

11. Secondary Outcome: Satisfaction of Diabetes Treatment Based on Diabetes Treatment Satisfaction Questionnaire Data
Description: The Diabetes Treatment Satisfaction Questionnaire allows to assess the degree of satisfaction with treatment for diabetes and its complications - retinopathy and nephropathy, how patients' satisfaction and perceived hyper- and hypoglycemia have changed compared to the initial period (before the treatment).
  The Diabetes Treatment Satisfaction Questionnaire contains six items scored on 7-point scales from +3 (equals "very satisfied") to -3 (equals "very dissatisfied"), with 0 (equals "no change"). These are summed to produce a total Treatment Satisfaction score. Two questions concerning "Perceived Hyperglycaemia" and "Perceived Hypoglycaemia" respectively, are calculated separately. According to these two items, low scores represent good perceived blood glucose control (+3 means "most of the time" of Hyperglycaemia or Hypoglycaemia whereas -3 means "none of the time" of Hyperglycaemia or Hypoglycaemia).
Time Frame: In 36 weeks of the treatment
Population: Intention-to-Treat set. 8 patients (6 in the Subetta group and 2 in the Placebo group) was excluded from the analysis due to lake of questionnaires.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Subetta | Placebo
Number analyzed (Participants) | 67 | 65
Scores on a scale
  Satisfaction | 9.8 (5.7) | 8.3 (6.1)
  Hyperglycemia | -1.1 (1.6) | -0.9 (1.7)
  Hypoglycemia | -1.1 (1.5) | -1.0 (1.6)
Statistical Analysis 1: Comparison: Subetta vs Placebo; Satisfaction; Test type: Superiority; p = 0.1577, t-test, 2 sided
Statistical Analysis 2: Comparison: Subetta vs Placebo; Hyperglycemia; Test type: Superiority; p = 0.5262, t-test, 2 sided
Statistical Analysis 3: Comparison: Subetta vs Placebo; Hypoglycemia; Test type: Superiority; p = 0.7417, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: Adverse/Serious adverse events were registered during 36 weeks of therapy and 30 days after the end of therapy.
Description: Adverse/Serious adverse events were registered in patients of the Full Analysis Set (n=148, Safety Population)
Arm/Group | Subetta | Placebo
Serious Adverse Events (participants affected / at risk) | 1/76 | 1/72
Other Adverse Events (participants affected / at risk) | 22/76 | 24/72
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Subetta (N=76) | Placebo (N=72)
Brain stem stroke (Nervous system disorders) | 1 | 0
Brain tumor NOS (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Subetta (N=76) | Placebo (N=72)
hypochromic anaemia (Blood and lymphatic system disorders) | 0 | 1
retinal angiopathy (Eye disorders) | 1 | 0
Diabetic edematous maculopathy (Eye disorders) | 1 | 0
Edema of the upper eyelid of the right eye (Eye disorders) | 1 | 0
duodenitis (Gastrointestinal disorders) | 0 | 1
burning tongue (Gastrointestinal disorders) | 0 | 1
epigastric burning (Gastrointestinal disorders) | 0 | 1
Periodic pain in the left hypochondrium (Gastrointestinal disorders) | 3 | 0
Periodic dull aching pain in the right hypochondrium (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 0
Drawing pains in the right hypochondrium (Gastrointestinal disorders) | 0 | 1
chronic gastritis (Gastrointestinal disorders) | 0 | 1
chronic colitis (Gastrointestinal disorders) | 0 | 1
Chronic parenchymal pancreatitis (Gastrointestinal disorders) | 1 | 1
Chronic hemorrhagic gastritis (Gastrointestinal disorders) | 1 | 0 — Chronic hemorrhagic gastritis, associated with Helicobacter, exacerbation
irritable bowel syndrome (Gastrointestinal disorders) | 1 | 0
Edema of the lower lip (Gastrointestinal disorders) | 1 | 0
esurience (General disorders) | 1 | 0
Complaints about general fatigue, a feeling of total severity and swelling (General disorders) | 1 | 0
Fatty liver hepatosis (Hepatobiliary disorders) | 1 | 1
allergic reaction (Immune system disorders) | 0 | 1
bilateral lacunar tonsillitis (Infections and infestations) | 1 | 0
Asymptomatic bacteriuria (Infections and infestations) | 0 | 1
upper respiratory infection (Infections and infestations) | 1 | 4
acute respiratory infection (Infections and infestations) | 4 | 10
upper respiratory tract infection (Infections and infestations) | 3 | 0
acute pneumonia (Infections and infestations) | 1 | 0
pulpitis (Infections and infestations) | 0 | 1
rhinitis (Infections and infestations) | 1 | 0
rhinosinusitis (Infections and infestations) | 1 | 0
Erysipelas of the right lower leg (Infections and infestations) | 0 | 1
pharyngitis (Infections and infestations) | 1 | 0
Fracture of radial head to the right (Injury, poisoning and procedural complications) | 0 | 1
Fracture of terminal phalanx of 5th toe of left foot (Injury, poisoning and procedural complications) | 0 | 1
Increased blood pressure (Investigations) | 4 | 2
rapid pulse (Investigations) | 0 | 1
Fasting hyperglycemia (Metabolism and nutrition disorders) | 1 | 0
hypercholesterinemia (Metabolism and nutrition disorders) | 0 | 1
Dyslipidemia, worsening (Metabolism and nutrition disorders) | 0 | 1
Increased appetite (Metabolism and nutrition disorders) | 0 | 1
Pain in the knee joints (Musculoskeletal and connective tissue disorders) | 1 | 0
melosalgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Pain in the lumbar spine (Musculoskeletal and connective tissue disorders) | 1 | 1
back pain (Musculoskeletal and connective tissue disorders) | 1 | 0
cervical vertebral osteochondrosis (Musculoskeletal and connective tissue disorders) | 1 | 0
headache (Nervous system disorders) | 0 | 1
occipital headache (Nervous system disorders) | 1 | 0
Diabetic distal sensory lower limb polyneuropathy, worsening (Nervous system disorders) | 1 | 0
Increased numbness in the fingers, feets (Nervous system disorders) | 1 | 0
Tingling in the region of the heart that occurs after excitement on a background of a stressful situ (Psychiatric disorders) | 1 | 0
Twitching of the right eye against a background of stress (Psychiatric disorders) | 0 | 1
phobic disorder (Psychiatric disorders) | 1 | 0
skin itch (Skin and subcutaneous tissue disorders) | 1 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 0
A papular rash in the area of the forearms, hands, right knee joint (Skin and subcutaneous tissue disorders) | 1 | 0
Urticaria on the extremities (Skin and subcutaneous tissue disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes